CLINICAL TRIAL: NCT05569161
Title: Prospective Multicentre Longitudinal Study to Evaluate the Safety and Clinical Radiological Outcomes in the First Two Years of the Ambrace Model Reverse Shoulder Arthroplasty.
Brief Title: To Evaluate the Safety and Clinical Radiological Outcomes in 2 Years of Embrance Model Reverse Shoulder Arthroplasty
Status: Recruiting | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Other Study IDs: PROTESISHOMBRO02
Record Dates: First submitted 2022-03-30; First posted 2022-10-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Implantation of a Reverse Shoulder Prosthesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The use of inverted prostheses to replace shoulder joints damaged by degenerative or traumatic processes has become widespread over the past three decades. Current designs, used correctly, can restore function and improve pain in the majority of patients in whom they are implanted.

The aim is to carry out a more detailed follow-up of the subjects who are implanted with this prosthetic model on a primary basis, analysing the clinical and radiological results and evaluating the presence of adverse effects of the prosthesis or short-term complications. For this purpose, subjects will be closely monitored for two years.

DETAILED DESCRIPTION:
The use of inverted prostheses to replace shoulder joints damaged by degenerative or traumatic processes has become widespread over the past three decades. Current designs, used correctly, can restore function and improve pain in the majority of patients in whom they are implanted.

However, there are complications associated with shoulder arthroplasty surgery, such as wear of the prosthetic components, infection, allergy to the prosthetic components, or failure to restore full shoulder function. The occurrence of these complications is affected by multiple factors dependent on the subject, the surgeon and/or the implant used.

ELIGIBILITY:
Inclusion Criteria:

* Patients who, after receiving information about the study design, the aims of the study, the possible risks that may arise from it and the fact that they may refuse to participate at any time, give their written consent to participate in the study.
* Be over 18 years of age.
* Have a shoulder joint disorder that is amenable to treatment with an Embrace reverse arthroplasty.
* Have a CT or MRI scan performed no more than 6 months prior to surgery.

Translated with www.DeepL.com/Translator (free version)

Exclusion Criteria:

* Patients who have undergone arthroplasty of any type on the ipsilateral shoulder.
* Patients with an active infection at any site at the time of shoulder surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital care consultations
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and the clinical and radiological outcome of Embrace primary reverse shoulder prostheses. | 24 months
  survival at 2-year follow-up with computerized tomografhic

SECONDARY OUTCOMES:
security | 24 months
  presence of possible adverse effects or complications, implant-related or not, including infection, mechanical complications of the implant, dislocation, fracture, loosening, readmission, reoperation or fracture.
efficiency | 24 months
  To evaluate the effect of the Embrace Reverse Embrace arthroplasty on postoperative pain and functional outcome. This is evaluate with computerized tomographic.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Ángel Ruiz Iban, Principal Investigator — IRYCIS. Hospital Universitario Ramón y Cajal. Madrid, Spain.
Locations (1):
- Miguel Ángel Ruiz Ibán, Madrid, Spain